CLINICAL TRIAL: NCT03558867
Title: Personalised Medicine in Prediabetes - Towards Preventing Diabetes in Individuals At Risk
Brief Title: Personalised Medicine in Pre-diabetes and Early Type 2 Diabetes
Acronym: PREDICT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Garvan Institute of Medical Research (Other)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SVH 17/080
Record Dates: First submitted 2018-06-05; First posted 2018-06-15 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2023-08

CONDITIONS: Pre Diabetes; Type 2 Diabetes Mellitus
Keywords: Pre Diabetes; Insulin resistance; Metformin; Gut microbiota; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Metformin; Diet, Healthy; Diet, Fat-Restricted; Diet

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin + Healthy diet (Placebo Comparator): Metformin (1500 mg/d, Extended Release) + Healthy, low fat diet
  Interventions: Drug: Metformin + Healthy diet
- Metformin + Personalized diet (Active Comparator): Metformin (1500 mg/d, Extended Release) + Personalized diet based on an algorithm developed at the Weizmann Institute of Science (Zeevi et al, Cell 2015)
  Interventions: Drug: Metformin + Personalized diet

INTERVENTIONS:
Drug: Metformin + Healthy diet — Metformin (1500 mg/d, Extended Release) + Healthy, low fat diet
  Other Names: Metformin + Healthy (low fat) diet
  Arms: Metformin + Healthy diet
Drug: Metformin + Personalized diet — Metformin (1500 mg/d, Extended Release) + Algorithm-based personalized diet
  Arms: Metformin + Personalized diet

SUMMARY:
Prediabetes is a common condition in overweight individuals affecting approximately 35% of American adults and 30% of Australian adults. Like diabetes, prediabetes is a serious risk factor for cardiovascular disease, eye, kidney and liver disease, and some types of cancer.

Appropriate blood glucose control is crucial in preventing pre-diabetes complications and onset of diabetes, yet clinical practice, backed by randomised trials, reports that many patients treated with standard dietary guidelines or with the first-line treatment of diabetes patients, metformin, do not improve blood glucose control sufficiently.

The overarching goal of the present project is to improve the efficacy of metformin mono-therapy in pre-diabetes and early type 2 diabetes.

DETAILED DESCRIPTION:
Prediabetes is common in overweight and obese individuals and, as with frank diabetes, it is a risk factor for cardiovascular disease, cognitive dysfunction, fatty liver, kidney, ophthalmic, renal and neuropathic disease, and cancer.

Effective management of dysglycemia in pre-diabetes and diabetes and prevention of diabetes in individuals at risk reduce the risk of organ damage and associated co-morbidities and improves the affected individuals' quality of life.

Metformin, an oral biguanide, is the first-line treatment of newly-diagnosed type 2 diabetes patients, and the pharmacological choice for preventing diabetes in individuals with pre-diabetes. Metformin is an ideal medication to initiate for diabetes prevention, due to its excellent safety profile (lack of hypoglycemia), neutral to marginally beneficial effect on body weight, evidence of cardio-protection, and low cost. However, clinical practice, backed by randomised clinical trials, suggests that metformin mono-therapy fails to achieve glycemic goals in 20-40% of type 2 diabetes patients and to prevent diabetes in approximately 20% of individuals with pre-diabetes.

While the mode of action of metformin is still being investigated, the liver and the gastrointestinal tract are thought to be the main targets responsible for the improvement in glycemia. An increasing body of evidence suggests that the gut microbiota play an important role in obesity, prediabetes and diabetes, and alterations in gut microbial composition have been described in individuals with type 2 diabetes and pre-diabetes. Interestingly, metformin-treated diabetes patients have a "healthier" gut microbial composition compared with treatment-naïve diabetes patients, and changes in gut microbial composition with metformin treatment has been suggested to contribute to the therapeutic effect of the medication.

Randomised, clinical study with parallel assignment and single-masking will be performed in treatment-naïve individuals with pre-diabetes or early type 2 diabetes (diagnosed in the last 6 months) aiming to compare the effect of metformin (extended release [XR]) 1500 mg/d administered with personalized diet (based on the Weizmann Institute Personalized Nutrition Project) or administered with a healthy (low fat) diet.

ELIGIBILITY:
Inclusion criteria:

* Individuals with pre-diabetes or newly-diagnosed (in the last 6 months) with type 2 diabetes, fulfilling the following criteria:
* Impaired fasting glucose (IFG, plasma glucose [PG]- 5.6 - 6.9 mmol/L, ±0.2 mmol/L) and/or impaired glucose tolerance (IGT, 2-h PG 7.8 - 11.0 mmol/L, ±0.2 mmol/L) with or without elevated HbA1c (up to 8.0 %).
* Willingness to provide written informed consent and willingness to participate and comply with the study.

Exclusion Criteria:

* Females planning a pregnancy during the course of the research or 3 months after completion of the research project.
* Patients with type 1 diabetes, chronically active inflammatory disease, neoplastic disease in the previous 3 years, chronic gastrointestinal disorders, including inflammatory bowel disease or celiac.
* Liver enzymes ALT and/or AST>3-times normal range limit.
* Abnormal renal function as measured by (eGFR<45 mL/min/1.73m^2).
* Individuals with a history of a psychological illness or condition that may interfere with the individual's ability to understand the requirements of the study.
* Normo-glycaemia.
* HbA1c>8.0%
* Cardiovascular event in the previous 6 months.
* Current or recent (within 24 months) treatment with a glucose lowering medication (i.e. GLP-1 receptor agonist, SGLT2 inhibitor, thiazolidinedione, sulfonylurea, DPP-4 inhibitor or insulin).
* Current or recent (within 3 months) treatment with metformin.
* Treatment with an oral steroid.
* Treatment with antibiotics/antifungal in the last 3 month.
* Treatment with immunosuppressive medications.
* Alcohol or substance abuse.
* Participants who had received an investigational new drug within the last 6 months.
* Participants involved in another clinical study.
* Participants who actively lose weight.
* Participants who had a bariatric surgery.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-07-23 (Actual)

PRIMARY OUTCOMES:
Mean change in glycated haemoglobin (HbA1C, %) from baseline | 6 months
  Difference in the reduction of HbA1C between the groups

SECONDARY OUTCOMES:
Total daily time of interstitial glucose levels below 7.8 mmol/L (140 mg/dL) | 6 months
  Difference in the time (minutes) per day with interstitial glucose measured below 7.8 mmol/L (140 mg/dL) between the groups
Glycaemic variability | 6 months
  Difference in the glycaemic variability as derived from CGM between the groups
Body weight | 6 months
  Difference in the magnitude of weight loss between the groups
Body fat mass | 6 months
  Difference in body fat mass composition as assessed using dual-energy X-ray absorptiometry (DXA) between the groups
Abdominal visceral fat volume | 6 months
  Difference in the abdominal visceral fat volume as assessed using DXA between the groups
Serum low-density lipoprotein (LDL)-cholesterol concentration | 6 months
  Difference in serum LDL-cholesterol between the groups
Serum high-density lipoprotein (HDL)-cholesterol concentration | 6 months
  Difference in serum HDL-cholesterol concentration between the groups
Serum triglycerides concentration | 6 months
  Difference in serum triglycerides between the groups
Blood pressure | 6 months
  Difference in diastolic and systolic blood pressure between the groups
Liver fat | 6 months
  Difference in liver fat measured by the Fibroscan's controlled attenuation parameter (CAP) function between the groups

OTHER OUTCOMES:
Gut microbiome (exploratory) | 6 months
  Difference in gut microbiome features between the groups

CONTACTS AND LOCATIONS:
Overall Officials: Dorit Samocha-Bonet, PhD, Principal Investigator — Garvan Institute of Medical Research; Jerry Greenfield, MD, PhD, Principal Investigator — Garvan Institute of Medical Research; Eran Elinav, MD, PhD, Principal Investigator — Weizmann Institute of Science; Eran Segal, PhD, Principal Investigator — Weizmann Institute of Science
Locations (1):
- Garvan Institute of Medical Research, Sydney, New South Wales, Australia

REFERENCES:
- [Derived] Htet TD, Godneva A, Liu Z, Chalmers E, Kolobkov D, Snaith JR, Richens R, Toth K, Danta M, Hng TM, Elinav E, Segal E, Greenfield JR, Samocha-Bonet D. Rationale and design of a randomised controlled trial testing the effect of personalised diet in individuals with pre-diabetes or type 2 diabetes mellitus treated with metformin. BMJ Open. 2020 Oct 10;10(10):e037859. doi: 10.1136/bmjopen-2020-037859. PMID 33040003
- See also: Study protocol paper — https://pubmed.ncbi.nlm.nih.gov/33040003/